CLINICAL TRIAL: NCT03623373
Title: A Pilot Study of Acalabrutinib With Bendamustine / Rituximab Followed by Cytarabine / Rituximab for Untreated Mantle Cell Lymphoma
Brief Title: Acalabrutinib With Bendamustine / Rituximab Followed by Cytarabine / Rituximab for Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201809111
Record Dates: First submitted 2018-07-26; First posted 2018-08-09 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab; acalabrutinib; Cytarabine; Leukapheresis; Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bendamustine/Rituximab/Acalabrutinib/Cytarabine (Experimental): * Patients will receive (6) 28 day cycles
  * Cycles 1-3 will consist of bendamustine on Days 1 and 2, rituximab on Day 1, and acalabrutinib twice per day (BID) on Days 1 through 28.
  * Cycles 4-6 will consist of rituximab on Day 1, cytarabine every 12 hours on Days 1 and 2, acalabrutinib BID on Days 1 through 7 and 22 through 28 (one week on, two weeks off, one week on), and growth factors as per institutional standard
  * After Cycle 6, patients will undergo leukapheresis
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Acalabrutinib; Drug: Cytarabine; Procedure: Leukapheresis; Procedure: Peripheral blood; Procedure: Oral rinse; Procedure: Bone marrow collection

INTERVENTIONS:
Drug: Bendamustine — Bendamustine will be administered at a dose of 90 mg/m^2 IV over 30 minutes on Days 1 and 2 of Cycles 1-3
  Other Names: Treanda; Bendeka
Drug: Rituximab — In Cycle 1, rituximab will be administered at a dose of 375 mg/m^2 IV on Day 1 or 2 at the investigator's discretion in order to reduce the risk of a first infusion reaction. Rituximab will be given on Day 1 of Cycles 1 through 6.
  Other Names: Rituxan; Rituxan Hycela
Drug: Acalabrutinib — The capsules should be swallowed intact with water and with or without food.
  Other Names: Calquence®
Drug: Cytarabine — On Days 1 and 2 of Cycles 4-6, following rituximab dosing, cytarabine will be administered IV every 12 hours for a total of 4 doses.
  Other Names: Cytosar-U
Procedure: Leukapheresis — Until collection of ≥ 2 x 106 CD34+ stem cells / kg
Procedure: Peripheral blood — -Baseline, end of Cycle 3, 4-6 weeks after Cycle 6 Day 1, and if the patient discontinues protocol therapy prior to completion of Cycle 6
Procedure: Oral rinse — -Baseline
Procedure: Bone marrow collection — -Bone marrow will be collected at baseline if the patient requires a marrow for staging purposes and at end of treatment if the patient requires a marrow for restaging.

SUMMARY:
This study is designed to evaluate the efficacy and safety of acalabrutinib plus bendamustine and rituximab followed by acalabrutinib plus cytarabine and rituximab in subjects with treatment naïve mantle cell lymphoma (MCL), as a preparation for a larger cooperative group trial with the goal of achieving a standard induction regimen for MCL in transplant eligible patients. The investigators hypothesize that the addition of acalabrutinib to BR/CR regimen will prove safe and increase the complete response (CR) rate as well as minimal residual disease (MRD) negativity pre-transplant, thus improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mantle cell lymphoma with documented expression of Cyclin D1 by immune-histochemical stains and/or t(11;14) by cytogenetics or FISH.
* Presence of evaluable disease by PET imaging per the Lugano classification.
* Eligible for autologous stem cell transplantation.
* Between 18 and 70 years of age, inclusive.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcL unless, in the opinion of the treating physician, neutropenia is due to splenomegaly or bone marrow involvement
  * Platelets ≥ 100,000/mcL unless, in the opinion of the treating physician, thrombocytopenia is due to splenomegaly or bone marrow involvement
  * Total bilirubin ≤ 2.0 x IULN and AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN except when, in the opinion of the treating physician, elevation is due to direct involvement of lymphoma (e.g. hepatic infiltration or biliary obstruction due to lymphoma) or Gilbert's disease
  * Creatinine ≤ IULN OR creatinine clearance ≥ 40 mL/min for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Any previous chemotherapy or radiation for mantle cell lymphoma. Short course of steroids for symptom relief prior to presentation is permissible.
* Symptomatic meningeal or parenchymal brain lymphoma.
* Prior exposure to a BTK inhibitor.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to acalabrutinib, rituximab, cytarabine, bendamustine, or other agents used in the study.
* Received a live virus vaccination within 28 days of first dose of study drug.
* Uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti-infective treatment within 2 weeks before first dose of study drug.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec at screening. Exception: subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll on study.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Active bleeding or history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of first dose of study drug.
* Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN. Exception: Subjects receiving warfarin are excluded; however, those receiving other anticoagulant therapy who have a higher INR/aPTT may be permitted to enroll to this study after discussion with the PI.
* Requires treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
* Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Subjects with serologic status reflecting active viral hepatitis B or C infection. Subjects who are hepatitis B core antibody positive but surface antigen negative will need negative polymerase chain reaction (PCR) prior to enrollment. Hepatitis B surface antigen positive or PCR positive patients will be excluded. Subjects who are hepatitis C antibody positive will need negative PCR prior to enrollment. Subjects with positive hepatitis C PCR will be excluded.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with acalabrutinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2025-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad S Kahl, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bendamustine/Rituximab/Acalabrutinib/Cytarabine
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine/Rituximab/Acalabrutinib/Cytarabine
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 57 [52 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Stem Cell Mobilization Success Rate With Cytarabine and Rituximab
Description: -Stem cell mobilization success is defined as a yield of >2x10^6 CD34+ stem cells/kg with a maximum of 5 courses of apheresis
Time Frame: Through 5 courses of apheresis (up to 5 days)
Population: 9 participants are not evaluable because they did not receive stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine/Rituximab/Acalabrutinib/Cytarabine
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Safety and Tolerability of Regimen in Subjects With MCL as Measured by Treatment Related Non-hematologic Toxicity of Grade 3 or Higher
Description: -Toxicity is measured using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: 30 days following completion of treatment (estimated to be 7 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine/Rituximab/Acalabrutinib/Cytarabine
Number analyzed (Participants) | 13
Participants
  Diarrhea | 1
  Infusion related reaction | 1
  Upper respiratory infection | 1
  Skin infection | 1
  Perirectal abscess | 1
  Peritoneal infection | 1
  Blood bilirubin increased | 1
  Ejection fraction decreased | 1
  Alanine aminotransferase increased | 1

3. Secondary Outcome: Overall Response Rate (ORR = Complete Response (CR) + Partial Response (PR)) of Subjects
Description: -For definitions of CR and PR please refer to the Recommendations for Initial Evaluation, Staging and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification
Time Frame: Through completion of treatment (estimated to be 6 months)
Population: 1 participant did not complete 2 cycles and was not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine/Rituximab/Acalabrutinib/Cytarabine
Number analyzed (Participants) | 12
Participants | 10

4. Secondary Outcome: Pre-transplant Complete Response Rate
Description: -For definitions of CR, please refer to the Recommendations for Initial Evaluation, Staging and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification
Time Frame: Through completion of treatment (estimated to be 6 months)
Population: 1 participant did not complete 2 cycles and was not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine/Rituximab/Acalabrutinib/Cytarabine
Number analyzed (Participants) | 12
Participants | 9

5. Secondary Outcome: Progression-free Survival (PFS)
Description: * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first
  * London Deauville score of 4 or 5 in individual target nodes/masses with an increase in intensity of uptake from the baseline and/or new FDG avid foci consistent with lymphoma at interim or end of treatment assessment; New FDG avid foci of extranodal disease consistent with lymphoma. If there is concern regarding the etiology of the new lesions, biopsy or interval scan may be considered; New or recurrent FDG avid foci in the bone marrow
Time Frame: Through 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival (OS)
Description: -OS=time from study registration until death from any cause
Time Frame: Through 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 30 days after the last dose of study treatment (approximately 7 months)
Arm/Group | Bendamustine/Rituximab/Acalabrutinib/Cytarabine
All-Cause Mortality (participants affected / at risk) | 3/13
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine/Rituximab/Acalabrutinib/Cytarabine (N=13)
Flu like symptoms (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Skin infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Infusion related reaction (General disorders) | 1
Retinal vein thrombosis (Eye disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Carcinoma of undetermined source (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine/Rituximab/Acalabrutinib/Cytarabine (N=13)
Anemia (Blood and lymphatic system disorders) | 12
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Stomach cramps (Gastrointestinal disorders) | 1
Tooth ache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Body aches (General disorders) | 2
Night sweats (General disorders) | 1
Chills (General disorders) | 1
Fever (General disorders) | 2
Edema limbs (General disorders) | 1
Malaise (General disorders) | 1
Fatigue (General disorders) | 9
Infusion related reaction (General disorders) | 5
Swelling (General disorders) | 1
Pain (General disorders) | 3
Allergic reaction (Immune system disorders) | 1
Upper respiratory infection (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Peritoneal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 3
Burning sensation at injection site (Injury, poisoning and procedural complications) | 1
Lymphocyte count decreased (Investigations) | 13
Blood bilirubin increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 13
Platelet count decreased (Investigations) | 13
Ejection fraction decreased (Investigations) | 1
White blood cell decreased (Investigations) | 13
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 4
Creatinine increased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Neuralgia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Keratosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Scalp scabs (Skin and subcutaneous tissue disorders) | 1
Diaphoresis (Skin and subcutaneous tissue disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 2
Hematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03623373/Prot_SAP_000.pdf